CLINICAL TRIAL: NCT03870464
Title: The Impact of Age and Comorbidity on Effect of Treatment, Adverse Effects and Quality of Life in Danish Lung Cancer Patients Receiving Immunotherapy
Brief Title: LIFE - Lung Cancer, Immunotherapy, Frailty, Effect
Status: Active, not recruiting | Type: Observational
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); University of Copenhagen (Other); Odense Patient Data Explorative Network (Other); Region of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: BBjornhart
Record Dates: First submitted 2019-03-01; First posted 2019-03-12 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Non-small Cell Lung Cancer; Quality of Life; Brain Metastases; Venous Thromboembolism
Keywords: non-small cell lung cancer; immunotherapy; checkpoint inhibition; biomarkers; quality of life; real life patients
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor-biopsies at baseline. Blood samples at baseline and consecutively
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective arm: Quality of Life questionnaires EORTC-QoL30 and Euro EQ-5D-5L questionnaires are distributed. Blood samples are collected consecutively during ICI and at a follow-up period of one year. CT-scans extended of thorax, abdomen and the lower extremities are performed at baseline and at 6 months. MRI scan of the brain screening for brain metastases. If brain metastases are diagnosed - the possibility of giving radiotherapy along the course of ICI is discussed with the patient. In case of brain metastases consecutive MRI scans of the brain will be performed in order to follow the course (natural or post-radiotherapy) of the disease.Prospective registration of irAEs are registered during ICI and for one year of follow-up.Enrolment period 1th of April 2018- 31th of April 2021.
  Interventions: Diagnostic Test: CT-scans extended; Diagnostic Test: MRI scan of the brain; Other: Prospective registration of irAEs; Behavioral: Quality of Life questionnaires

INTERVENTIONS:
Diagnostic Test: CT-scans extended — CT scans of thorax, abdomen and lower extremities are performed - screening for venous trombolisms at baseline and at 6 months in each patient. If VTE is diagnosed, medications according to guidelines will be administered.
Diagnostic Test: MRI scan of the brain — MRI scan of the brain screening for brain metastases. If brain metastases are diagnosed - the possibility of giving radiotherapy along the course of ICI is discussed with the patient. In case of brain metastases consecutive MRI scans of the brain will be performed in order to follow the course (natural or post-radiotherapy) of the disease.
Other: Prospective registration of irAEs — irAEs are registered according to Common Terminology Criteria for Adverse Events version 4.0 by a medical doctor or trained experienced clinical nurse.
Behavioral: Quality of Life questionnaires — Participants fill out two Quality of Life questionnaires. The European Organization of Research and Treatment of Cancer, Quality of Life -30 questionnaire (EORTC QoL-30) and the European Questionnaire - 5 dimensions-5-level questionnaire (Euro EQ-5D-5L).

SUMMARY:
The LIFE study (Lung cancer, Immunotherapy, Frailty, Effect) is investigating the unselected 'real life' non-small cell lung cancer (NSCLC) population treated with immune checkpoint inhibition.

DETAILED DESCRIPTION:
The era of immune checkpoint inhibition (ICI) has changed the treatment regimen for incurable non-small cell lung cancer. With that the hope of a more long-term survival has been introduced. ICI is given as standard therapy for selected NSCLC patients with incurable advanced or metastatic (stage IV) disease. For this group of patients clinical trial reports present a 3 year overall survival rate of around 30%. Checkpoint inhibition is also known as programmed death 1 (PD-1) or programmed death-ligand 1 (PD-L1) inhibitors and the PD-L1 tumor proportion score is currently the only clinically applicable biomarker used for this patient selection. New prognostic and predictive biomarkers are therefore warranted.The real life unselected NSCLC patient eligible for treatment with immunotherapy (check point inhibition) may be both older, with more comorbidity, more widespread disease and in poorer performance status than patients treated in clinical phase III trials. In this prospective single center study, clinical patient data, peripheral blood and baseline pre-treatment tumor biopsies are collected from NSCLC patients treated in any given treatment line with nivolumab, pembrolizumab or atezolizumab. Besides baseline samples consecutive blood samples will be collected for cytokine profiling and measurement of circulating tumor DNA (ctDNA) and micro RNA analysis. Baseline MRI of the brain screening for brain metastases and an extended CT-scan of thorax, abdomen and the lower extremities will be performed screening for venous thromboembolism (VTE). This along with comorbidity screening tools and quality of life assessments will provide detailed mapping of both patient and disease characteristics of potentially more frail patients including those with untreated brain metastases. By also registering immune related adverse events (irAE) prospectively in this study and doing additional blood samples in case of grade 3-4 toxicity, identification of biomarkers as predictors for effect and toxicity is durable. Hopefully this will contribute to more optimized treatment courses for those NSCLC patients to come.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Stage IV NSCLC or recurrent NSCLC.
* Squamous or non-squamous histology
* Any treatment-line - Independent of prior treatment
* Candidate for checkpoint inhibitor (PD-1/PD-L1 targeting agents) immunotherapy
* No previously known allergy to PD-1/PD-L1 targeting agents.
* Able to give written consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 150 patients with incurable advanced (stage III A-C) or metastatic (stage IV) non-small cell lung cancer eligible for treatment with ICI at a Danish Hospital (Odense, Denmark). All possible treatment lines are allowed. ICI administered as nivolumab, pembrolizumab or atezolisumab.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with CTCAE 4.0 toxicity registered Immune related autoimmune events (irAE). | ICI will be given for a maximum of 24 months, and irAE registered up till one year post ICI treatment, which is anticipated to be within 4 years after of start inclusion.
  Number of patients with CTCAE 4.0 toxicity registered according to age, comorbidity and predictive biomarkers.
Effect of checkpoint inhibition | ICI will be given for a maximum of 24 months, and follow-up is a maximum of one year post ICI, therefore is anticipated to be compleated within 4 years after start of inclusion.
  Effect of ICI by calculating patients' overall median survival time.
Potential biomarkers for patient outcome including cDNA, mRNA and coagulation markers. | ICI will be given for a maximum of 24 months, and during follow-ip of one year post ICI treatment. Therefore it is anticipated to be compleated within 4 years after start inclusion
  Investigations of blood samples stored in a biobank. These include cDNA, mRNA, acute phase reactants, markers of coagulation.
Effect of checkpoint inhibition | ICI will be given for a maximum of 24 months, and during follow-ip of one year post ICI treatment. Therefore it is anticipated to be compleated within 4 years after start inclusion.
  Effect of ICI by calculating patients' median progression free survival time.
Best response of checkpoint inhibition | ICI will be given for a maximum of 24 months, and during follow-ip of one year post ICI treatment. Therefore it is anticipated to be compleated within 4 years after start inclusion.
  Best response during ICI in patients, defined as radiologic response rates using CT evaluations (Recist 1.1 criteria) combined with clinical status during ICI.

SECONDARY OUTCOMES:
Registration of venous thromboembolism (VTE) during treatment with ICI. | ICI will be given for a maximum of 24 months, which is anticipated to be within 4 years after start inclusion
  Registration of VTE during treatment with ICI using expanded CT scans at baseline/6 months.
The Quality of Life in patients at baseline and at follow-up using EORTC QoL-30. | ICI will be given for a maximum of 24 months, and the follow-up period is one year, therefore completion is anticipated to be within 4 years after start inclusion.
  Questionnaires of EORTC-Quality of Life-30 (EORTC QoL-30).
The Quality of Life in patients at baseline and at follow-up using European EQ-5D-5L). | ICI will be given for a maximum of 24 months, and the follow-up period is one year, therefore completion is anticipated to be within 4 years after start inclusion.
  Evaluating Quality of Life using the European Quality of life - 5 Dimensions - 5 Levels questionnarie (Euro EQ-5D-5L) at baseline, during treatment and at follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte Bjørnhart, MD, Principal Investigator — University of Southern Denmark
Locations (1):
- Department of Oncology, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided